CLINICAL TRIAL: NCT03035851
Title: Aerobic Exercise for Older Adults at Increased Risk of Alzheimer's Disease and Related Dementias: Harnessing Translational Physiology
Brief Title: Aerobic Exercise for Older Adults at Increased Risk of Alzheimer's Disease and Related Dementias
Acronym: BIMII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marc Poulin, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REB 16-1199
Record Dates: First submitted 2016-12-22; First posted 2017-01-30 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer Disease; Dementia; Exercise; Physical Activity; Brain blood flow; Cognition; Fitness
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental): Participants will take part in a supervised 6-month-long aerobic (walk/jog) training program held 3 days/week. Each session will include a 5-min warm-up, 20-40 min of aerobic exercise (walking, jogging), 5-min cool-down, and stretching. Exercise prescriptions will follow current principles and guidelines established by ACSM/AHA, including sufficient warm-up, cool-down, and ongoing provision of safety precautions/exercise tips. As participants progress, the duration of aerobic exercise will increase from 20 (month 1) to 30 (months 2-3) and 40 min (months 4-6), with proportional increases to warm-up and cool-down periods. Exercise intensity will be based on individual maximal oxygen uptake (VO2 max), measured at baseline. Intensity will build from 30-45% (months 1-3) to mitigate the risk of injury and will progress to 60-70% (months 4-6) heart rate reserve (HRR).
  Interventions: Behavioral: Aerobic exercise
- Stretch and Strength (Other): A control group will meet on a similar schedule as the exercise group for sessions on stretching and toning but without aerobic exercise. Based on prior RCTs of similar interventions the investigators expect this control to be ineffective or minimally effective, but anticipate that it will increase participant enthusiasm and retention. All assessments will be conducted in this arm.
  Interventions: Behavioral: Stretch and Strength

INTERVENTIONS:
Behavioral: Aerobic exercise
  Arms: Aerobic exercise
Behavioral: Stretch and Strength
  Arms: Stretch and Strength

SUMMARY:
The estimated annual cost of dementia in Canada is $15 billion, with a projected cumulative economic burden of $800 billion by 2038. Effective prevention of dementia at a population level will need to include lifestyle factors such as promoting higher levels of physical activity. Physical inactivity is a modifiable risk factor for Alzheimer disease (AD) and cognitive decline, but the mechanisms by which physical activity exerts its protective effect on the brain remain unknown. Motivated by the need to develop strategies to prevent and treat AD and related dementias (ADRD), the investigators' overall research goal is to discover why the aging brain develops ADRD. To achieve this goal the investigators adopt a translational physiology approach (i.e., study of physiology from molecule/cell to population) to investigate how exercise improves cognitive performance, and the underlying mechanisms by which exercise prevents and/or slows down age-related declines in brain health and cognition. This approach allows the investigators to determine how physiological function is related to ADRD, with important implications for health. The investigators' prior work demonstrated a significant relationship between fitness, vascular regulation and cognition in older adults free of overt disease. These findings have implications for vascular cognitive impairment and ADRD, in which hypoperfusion and dysregulation of cerebral blood flow are thought to be important pathophysiological factors. The investigators' central hypothesis is that regular aerobic exercise mitigates age-related decreases in vascular function and cerebrovascular reserve, which in turn benefits cognition. Work by the investigators and others has provided the necessary data justifying a randomized controlled trial to evaluate the role of exercise in the prevention of ADRD.

The investigators are well equipped to undertake this trial; the investigators have dedicated institutional support and necessary expertise in vascular regulation, cognition, aging, neuroimaging and genetics.

The overall objective of this proposal is to test an exercise intervention for secondary prevention of ADRD in adults between 50 and 80 years old who are at increased risk for ADRD (with memory impairment symptoms but without dementia). The rationale for this trial is the urgent need for dementia prevention: an exercise intervention, which harnesses a translational physiology framework, holds such promise. The investigators will conduct this trial to determine the effects of aerobic exercise on the development of age-associated cognitive decline and dementia. The exercise intervention is designed with input from Alberta Health Services, the universal healthcare provider for Albertans, so that the intervention can be readily adopted into clinical practice if this trial is successful. The trial will address three specific aims.

SPECIFIC AIM 1: Determine the independent effect of exercise on cognitive performance in previously inactive older adults at increased risk of ADRD. The investigators hypothesize that participants randomized to our six-month aerobic exercise intervention will perform better on cognitive tests, compared to control participants randomized to a stretching-toning exercise group.

SPECIFIC AIM 2: Determine underlying biological mechanisms that influence cognitive performance after exercise training. The investigators hypothesize that exercise improves cognition due to changes at molecular/cellular (biomarkers), vascular (cerebral blood flow, cerebrovascular reserve), anatomical and functional (neuroimaging), and behavioural (sleep quality) levels. Further, the investigators hypothesize that ADRD-specific genetic risk scores, reflective of targeted genetic variants, moderate exercise-related cognitive and brain outcomes.

SPECIFIC AIM 3: Determine the extent to which changes in cognition, resting cerebral blood flow and cerebrovascular reserve persist 12 months after participants complete a 6-month exercise training intervention. The investigators hypothesize that the effects of improved aerobic fitness will be maintained over time as a function of persistent lifestyle changes and behavioural support programs. This trial will provide evidence needed to make clinical recommendations for exercise programs in adults at risk for ADRD, with the goal of preventing dementia. Given the investigators' extensive stakeholder input, this intervention will be easily translated to other jurisdictions. This research into the mechanisms of effect for exercise will identify patient subgroups most likely to benefit, surrogate outcome markers for use in future trials to refine intervention dose/duration, and new therapeutic targets for future interventions.

ELIGIBILITY:
Inclusion Criteria:

* inactive men and women aged 50-80 years (inclusive) with subjective cognitive symptoms but no dementia who have one or more vascular risk factors (see below) for ADRD;
* Inactivity will be assessed with a physical activity questionnaire and defined as engagement in <3 sessions/week of 20 min or more of vigorous exercise;
* Subjective cognitive symptoms will be self-reported using the MAC-Q Memory Complaint Questionnaire, recently validated as a measure of subjective memory complaints in healthy elderly subjects, in patients with mild cognitive impairment, and in relation to AD biomarkers; participants with a score of ≥25 will be considered eligible.
* Vascular risk factors for ADRD including the following:
* history of hypertension;
* diabetes mellitus;
* obesity (body mass index (BMI) <40 kg/m2)
* elevated cholesterol;
* currently smoking;
* past history of coronary artery disease without recent (<5 years) symptoms.

Participants must provide a completed PAR-Q+ form (www.csep.ca), the standard method of obtaining physician approval for participation in an exercise program. For participants without a family doctor to provide this form, we will provide information on how to find a family doctor.

Exclusion Criteria:

* diagnosis of a developmental handicap;
* history of dementia (DSM-V criteria)**;
* terminal illness (life expectancy < 1 year)
* not fluent in verbal and written English;
* history of stroke;
* currently participating in another trial;
* comorbid medical or neurological illnesses (e.g., multiple sclerosis) that would confound cognitive assessments or make trial completion unlikely (in the site investigator's opinion);
* contraindication for the intervention;
* contraindication for an MRI exam.
* **Existing or suspected dementia will be identified by medical history, cognitive impairment on the Telephone Interview for Cognitive Status (TICS-modified; score≤ 20), or impaired Instrumental Activities of Daily Living (IADL) - a response of needs assistance or dependent due to cognitive impairments on any item on the Lawton scale.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2017-01; Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition Assessed by Neuropsychological Test Battery | Measured at baseline, exercise intervention completion (6 months) and follow-up (18 months)

SECONDARY OUTCOMES:
Change in Cerebral Blood Flow Assessed by Transcranial Doppler Ultrasound | Participants will be assessed at baseline, at the completion of the intervention (6 months) and at follow-up (18 months) phases of the study.
Change in Maximal Oxygen Uptake (VO2max) Assessed by Metabolic Cart | Participants will be assessed at baseline, at the completion of the intervention (6 months) and at follow-up (18 months) phases of the study.
  The change in aerobic fitness will be assessed by VO2max, determined by cardiopulmonary stress testing.
Change in Blood Biomarkers Assessed by Elisa Assays | Participants will be assessed at baseline, at the completion of the intervention (6 months) and at follow-up (18 months) phases of the study.
  blood sampling and analyses of the selected markers (e.g., neurotrophins, cytokines, inflammatory markers, cortisol, oxidative stress, NO and antioxidants).
Change in Risk/protective factors Assessed by Questionnaires | Participants will be assessed at baseline, at the completion of the intervention (6 months) and at follow-up (18 months) phases of the study.
  Measures include changes in dietary intake, food frequency, supplement intake, physical activity, cognitive activities, mood changes, social support and engagement.
Change in Brain Structure and Function Assessed by Neuroimaging Modalities | Participants will be assessed at baseline, at the completion of the intervention (6 months) and at follow-up (18 months) phases of the study.
Change in Sleep Quality Assessed by Polysomnography, Actigraphy and Questionnaires | Participants will be assessed at baseline, at the completion of the intervention (6 months) and at follow-up (18 months) phases of the study.
Change in Health behaviour with appropriate support strategies | Participants will be assessed at 6, 12 and 18 months.
  The investigators will assess whether, in the 12-month period following the 6-month exercise intervention, individually-tailored, telephone support for home-based exercise improves adherence and sustains the beneficial effects of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Poulin, PhD, DPhil, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Kruger RL, Clark CM, Dyck AM, Anderson TJ, Clement F, Hanly PJ, Hanson HM, Hill MD, Hogan DB, Holroyd-Leduc J, Longman RS, McDonough M, Pike GB, Rawling JM, Sajobi T, Poulin MJ. The Brain in Motion II Study: study protocol for a randomized controlled trial of an aerobic exercise intervention for older adults at increased risk of dementia. Trials. 2021 Jun 14;22(1):394. doi: 10.1186/s13063-021-05336-z. PMID 34127029